CLINICAL TRIAL: NCT01747902
Title: Biceps Tenodesis Versus Tenotomy in the Treatment of Lesions of the Long Head of Biceps Brachii: a Randomized Controlled Trial
Brief Title: Biceps Tenodesis Versus Tenotomy
Acronym: BicepsTvsT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panam Clinic (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Principal Investigator, Peter MacDonald, Department Head, Orthopaedics, Panam Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2012:113
Record Dates: First submitted 2012-12-05; First posted 2012-12-12 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Rotator Cuff Tear; Long Head of Biceps Brachii Lesions
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biceps tenodesis (Other): The biceps tenodesis group will have their bicep detached and then re-inserted onto the shoulder.
  Interventions: Procedure: Biceps Tenodesis
- Biceps Tenotomy (Other): The biceps tenotomy group will have their bicep treated by detaching the tendon from the shoulder.
  Interventions: Procedure: Biceps Tenotomy

INTERVENTIONS:
Procedure: Biceps Tenotomy — The biceps tenotomy group will have their bicep treated by detaching the tendon from the shoulder.
  Arms: Biceps Tenotomy
Procedure: Biceps Tenodesis — The biceps tenodesis group will have their bicep detached and then re-inserted onto the shoulder.
  Arms: Biceps tenodesis

SUMMARY:
The long head of biceps brachii tendon has been known to be a pain generator and a common cause of shoulder pain and dysfunction in patients with rotator cuff pathology. Both biceps tenotomy and tenodesis have been shown to produce comparable results, but there is no consensus to date due to a lack of level I evidence. The aim of this prospective, randomized, clinical trial is to compare subjective patient-reported outcomes and objective clinical results between biceps tenotomy and biceps tenodesis for treating lesions of the long head of the biceps brachii.

DETAILED DESCRIPTION:
Methodology

Patients will be screened in clinic and, if deemed appropriate for the study, will be approached by the research coordinator who will review the study and provide the opportunity for consenting to participate. The surgical procedure will be performed using standard arthroscopic technique and patients will be randomized intra-operatively via computer randomization when a biceps tendon lesion is confirmed. The type of anchor for the tenodesis, whether bioabsorbable or metal, and the manufacture of the anchor used is at the discretion of the surgeon. Duration of the surgery will be between 60-120 minutes.

Surgical Technique

The technique can be done using a biceps groove or a subpectoral level of fixation depending on surgeon preference. Shoulder arthroscopy is conducted in the lateral decubitus or beach chair position. Diagnostic arthroscopy is performed using a standard posterior portal and the biceps tendon is assessed with an arthroscopic probe using a standard anterior interval portal. Once study eligibility was confirmed via identification of tearing or degeneration of the long head of biceps, the patient was randomized to undergo either tenodesis or tenotomy.

For patients who undergo biceps tenotomy the long head of biceps tendon is detached from its proximal anchor to the superior labrum using an arthroscopic biter, an electrothermal device, or a scalpel based on individual surgeon preference.

For those patients undergoing biceps tenodesis, the tendon is tagged with a monofilament suture prior to detaching it from its superior labral attachment. The long head of biceps is then mobilized arthroscopically, and retrieved through an incision either in the groove (which is opened arthroscopically in the subacromial space) or at the inferior border of the pectoralis major tendon. A No. 2 non-absorbable suture is whip-stitched at the appropriate length. The remainder of the biceps tendon is excised and the anterior cortex of the proximal humerus is prepared using a cannulated reamer inserted into the bicipital groove. One suture limb is then passed through an appropriate size interference screw and the tendon is placed within the reamed tunnel. The screw is then advanced until it is flush with bone..

Once the long head of biceps tendon pathology had been addressed, the scope is switched to a standard lateral portal to assess subacromial pathology and the rotator cuff. Subacromial decompression is performed using a cutting block technique if required, and the rotator cuff is repaired if necessary using standard anterolateral and posterolateral accessory portals based on tear configuration.

Post-operative Care and Physiotherapy

Postoperative care and immobilization are identical for the two groups and consist of the use of an immobilizer for 4-6 weeks. Patients are allowed to remove the immobilizer for activities of daily living in which the arm is not abducted and does not externally rotate beyond neutral. Active range of motion is started at 4-6 weeks and resistance exercises are begun when maximal range of motion has been achieved. No at-risk work activities or sports are allowed for six months.

Data Analysis

The primary analysis involves a comparison of the mean ASES scores between the two surgical treatment groups on an intention to treat basis. This analysis is a two sample independent t-test to assess whether there is a statistically significant difference between groups for the mean ASES scores at baseline and each follow-up appointment up to two years. Repeated measures ANOVAs will be used to determine the effect of surgery from baseline to two years post-surgery (i.e. pre-operatively, 3, 6, and 12, and 24 month follow-ups) on ASES scores for each group. The 5% significance level is employed. The underlying assumption for the ASES score data is that there is a normal distribution. If the sample distribution is determined to depart from normal, then a Wilcoxon rank sum test with Bonferroni correction will be performed. The secondary analysis involves a comparison of the secondary outcome measures between the two surgical treatment groups. The elbow strength findings will be analyzed for differences between the two groups at each time point up to 2 years. Repeated measures ANOVAs will be used to determine the effect of surgery from baseline to two years post-surgery (i.e. pre-operatively, 3, 6, and 12, and 24 month follow-ups) on ASES and elbow strength for each group. Nominal demographic data will be compared using the chi-squared test, while ordinal data will be compared using a t-test.

Significance of the Proposed Research

Arthroscopic treatment of lesions of the long head of the biceps tendon, whether tenodesis or tenotomy, has shown consistently favourable results. This trial is necessary both to provide optimal care of our patients, and to do so in a fiscally responsible fashion as the biceps tenodesis procedure has potential cost implications related to additional surgical time and anchor requirements. The results of the trial will provide valuable information regarding the management of lesions of the long head of the biceps tendon. The data obtained from quality of life measurements and physical exam will enable the authors to make recommendations that will lead to maximizing shoulder function and quality of life in patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Must benefit from arthroscopic rotator cuff surgery and inta-operative findings must confirm a lesion of the long head of biceps tendon

Exclusion Criteria:

* Any significant comorbidities including previous surgery on affected shoulder
* Active worker's compensation claims
* Active joint or systemic infection, significant muscle paralysis, Charcot's arthropathy
* Significant medical comorbidity that could alter the effectiveness of the surgical intervention (e.g., Cervical radiculopathy, polymyalgia rheumatica)
* Major medical illness (life expectancy less then one year or unacceptably high operative risk)
* Inability to speak or read English/French
* Psychiatric illness that precludes informed consent
* Unwillingness to be followed for 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-01; Primary Completion 2018-04 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
American Should and Elbow Society (ASES) | 24 months

SECONDARY OUTCOMES:
Operative Time | 24 months
  Total operative time in tenodesis vs. tenotomy procedures
Incidence of Revision | 24 months
  How many of each group will return for some form of surgical revision.
Complications | 24 months
  Surgical complications present in both tenotomy and tenodesis groups.
Magnetic Resonance Imaging (MRI) | 24 months
  To be obtained at one year post-operatively to assess the integrity of the tenodesis procedure, and the amount of tendon retraction in the tenotomy group.
Strength | 24 months
  Shoulder strength
Range of Motion | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter MacDonald, MD FRCSC, Principal Investigator — Pan Am Clinic
Locations (1):
- Pan Am Clinic, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Friedman DJ, Dunn JC, Higgins LD, Warner JJ. Proximal biceps tendon: injuries and management. Sports Med Arthrosc Rev. 2008 Sep;16(3):162-9. doi: 10.1097/JSA.0b013e318184f549. PMID 18703976
- [Background] Szabo I, Boileau P, Walch G. The proximal biceps as a pain generator and results of tenotomy. Sports Med Arthrosc Rev. 2008 Sep;16(3):180-6. doi: 10.1097/JSA.0b013e3181824f1e. PMID 18703979
- [Background] Frost A, Zafar MS, Maffulli N. Tenotomy versus tenodesis in the management of pathologic lesions of the tendon of the long head of the biceps brachii. Am J Sports Med. 2009 Apr;37(4):828-33. doi: 10.1177/0363546508322179. Epub 2008 Sep 1. PMID 18762669
- [Background] Koh KH, Ahn JH, Kim SM, Yoo JC. Treatment of biceps tendon lesions in the setting of rotator cuff tears: prospective cohort study of tenotomy versus tenodesis. Am J Sports Med. 2010 Aug;38(8):1584-90. doi: 10.1177/0363546510364053. Epub 2010 Jun 15. PMID 20551285
- [Background] Kelly AM, Drakos MC, Fealy S, Taylor SA, O'Brien SJ. Arthroscopic release of the long head of the biceps tendon: functional outcome and clinical results. Am J Sports Med. 2005 Feb;33(2):208-13. doi: 10.1177/0363546504269555. PMID 15701606
- [Background] Boileau P, Krishnan SG, Coste JS, Walch G. Arthroscopic biceps tenodesis: a new technique using bioabsorbable interference screw fixation. Arthroscopy. 2002 Nov-Dec;18(9):1002-12. doi: 10.1053/jars.2002.36488. PMID 12426544
- [Background] Walch G, Edwards TB, Boulahia A, Nove-Josserand L, Neyton L, Szabo I. Arthroscopic tenotomy of the long head of the biceps in the treatment of rotator cuff tears: clinical and radiographic results of 307 cases. J Shoulder Elbow Surg. 2005 May-Jun;14(3):238-46. doi: 10.1016/j.jse.2004.07.008. PMID 15889020
- [Background] Boileau P, Baque F, Valerio L, Ahrens P, Chuinard C, Trojani C. Isolated arthroscopic biceps tenotomy or tenodesis improves symptoms in patients with massive irreparable rotator cuff tears. J Bone Joint Surg Am. 2007 Apr;89(4):747-57. doi: 10.2106/JBJS.E.01097. PMID 17403796
- [Background] Edwards TB, Walch G, Sirveaux F, Mole D, Nove-Josserand L, Boulahia A, Neyton L, Szabo I, Lindgren B, O'Connor DP. Repair of tears of the subscapularis. Surgical technique. J Bone Joint Surg Am. 2006 Mar;88 Suppl 1 Pt 1:1-10. doi: 10.2106/JBJS.E.00842. PMID 16510795
- [Background] Osbahr DC, Diamond AB, Speer KP. The cosmetic appearance of the biceps muscle after long-head tenotomy versus tenodesis. Arthroscopy. 2002 May-Jun;18(5):483-7. doi: 10.1053/jars.2002.32233. PMID 11987057
- [Background] Slenker NR, Lawson K, Ciccotti MG, Dodson CC, Cohen SB. Biceps tenotomy versus tenodesis: clinical outcomes. Arthroscopy. 2012 Apr;28(4):576-82. doi: 10.1016/j.arthro.2011.10.017. Epub 2012 Jan 28. PMID 22284407
- [Background] Duff SJ, Campbell PT. Patient acceptance of long head of biceps brachii tenotomy. J Shoulder Elbow Surg. 2012 Jan;21(1):61-5. doi: 10.1016/j.jse.2011.01.014. Epub 2011 Mar 30. PMID 21454097
- [Background] Wolf RS, Zheng N, Weichel D. Long head biceps tenotomy versus tenodesis: a cadaveric biomechanical analysis. Arthroscopy. 2005 Feb;21(2):182-5. doi: 10.1016/j.arthro.2004.10.014. PMID 15689867
- [Background] Shank JR, Singleton SB, Braun S, Kissenberth MJ, Ramappa A, Ellis H, Decker MJ, Hawkins RJ, Torry MR. A comparison of forearm supination and elbow flexion strength in patients with long head of the biceps tenotomy or tenodesis. Arthroscopy. 2011 Jan;27(1):9-16. doi: 10.1016/j.arthro.2010.06.022. Epub 2010 Oct 29. PMID 21035992
- [Background] Richards RR, An KN, Bigliani LU, Friedman RJ, Gartsman GM, Gristina AG, Iannotti JP, Mow VC, Sidles JA, Zuckerman JD. A standardized method for the assessment of shoulder function. J Shoulder Elbow Surg. 1994 Nov;3(6):347-52. doi: 10.1016/S1058-2746(09)80019-0. Epub 2009 Feb 13. PMID 22958838
- [Background] Michener LA, McClure PW, Sennett BJ. American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form, patient self-report section: reliability, validity, and responsiveness. J Shoulder Elbow Surg. 2002 Nov-Dec;11(6):587-94. doi: 10.1067/mse.2002.127096. PMID 12469084
- [Derived] MacDonald P, Verhulst F, McRae S, Old J, Stranges G, Dubberley J, Mascarenhas R, Koenig J, Leiter J, Nassar M, Lapner P. Biceps Tenodesis Versus Tenotomy in the Treatment of Lesions of the Long Head of the Biceps Tendon in Patients Undergoing Arthroscopic Shoulder Surgery: A Prospective Double-Blinded Randomized Controlled Trial. Am J Sports Med. 2020 May;48(6):1439-1449. doi: 10.1177/0363546520912212. Epub 2020 Mar 30. PMID 32223645